CLINICAL TRIAL: NCT05249205
Title: The Effect of Training Frequency on Improvements in Maximal Aerobic Capacity With Reduced-exertion High-intensity Interval Training (REHIT)
Brief Title: The Effect of Training Frequency on Improvements in VO2max With REHIT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues with key equipment
Sponsor: University of Stirling (Other)
Collaborators: Swansea University (Other); University of Worcester (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal investigator, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NICR4056
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: General Health
Keywords: Reduced-exertion high-intensity interval training; REHIT; Training frequency; Fitness

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: The nature of the intervention does not allow for blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the control group will be asked to maintain their regular lifestyle for the duration of the study. They will not receive an intervention.
- REHIT1 (Experimental): Participants in the REHIT1 group will perform a single REHIT session per week for 6 weeks.
  Interventions: Behavioral: REHIT1
- REHIT2 (Experimental): Participants in the REHIT2 group will perform 2 REHIT sessions per week for 6 weeks.
  Interventions: Behavioral: REHIT2

INTERVENTIONS:
Behavioral: REHIT1 — This intervention involves a single REHIT exercise session per week. REHIT involves 10 minutes of unloaded cycling on a stationary bike interspersed with two 20-second 'all-out' cycle sprints against a resistance equivalent to 7.5% of body mass.
  Other Names: Reduced-exertion high-intensity interval training / single session per week
  Arms: REHIT1
Behavioral: REHIT2 — This intervention is the same as that for the REHIT1 intervention, but with 2 sessions per week instead of 1.
  Other Names: Reduced-exertion high-intensity interval training / 2 sessions per week
  Arms: REHIT2

SUMMARY:
Many people do not manage to do the recommended amount of physical activity for improving general health and wellbeing, and a common reason for this is lack of time. Sprint interval training (SIT) has been suggested to be a time-efficient alternative to current exercise recommendations, but most SIT protocols are not actually as time-efficient as claimed. However, it has previously been shown that the training time commitment of common SIT protocols can be substantially reduced while remaining effective at improving key health markers such as aerobic fitness, insulin function and blood pressure. For example, the reduced-exertion high-intensity interval training (REHIT) protocol consists of two 20-second 'all-out' cycle sprints within a 10-minute low-intensity exercise session. There is some evidence that REHIT is just as effective at improving aerobic fitness with 2 exercise sessions per week compared to 3 or 4 sessions. However, it remains unknown if improvements in aerobic fitness are reduced if just a single REHIT session is performed each week. Therefore, the aim of the present study is to compare improvements in aerobic fitness levels between a control group (no training intervention), a group performing a single REHIT session per week, and a group performing 2 REHIT sessions per week.

DETAILED DESCRIPTION:
Up to 45 apparently healthy participants will be recruited at multiple sites. Eligible participants will complete a fitness test to measure pre-training maximal aerobic capacity (V̇O2max). Participants will start cycling on a stationary bike at a low intensity (30 W). The intensity will increase by 1 W every 3 seconds until volitional exhaustion or an inability to maintain a pedalling frequency of >60 rpm. Expired O2 and CO2 will be continuously measured breath-by-breath using an online gas analyser. V̇O2max will be determined as the highest value for a 15-breath rolling average of V̇O2. V̇O2max will be accepted if at least 2 of the following criteria are met: volitional exhaustion / inability to maintain a pedal frequency of 60 rpm, RER>1.10, a plateau in V̇O2, and/or heart rate within 10 bpm of the age predicted maximum (220-age).

Participants will then be randomised into one of 3 groups, performing either 1 or 2 REHIT training sessions per week, or no training intervention (control group). Randomisation will be performed using the sealed envelope method. Participants in the control group will be asked to maintain their regular lifestyle for 6 weeks. Participants in the training groups will perform 6 weeks of REHIT. Each REHIT session involves 10 min of unloaded pedalling interspersed with 2 all-out cycle sprints against a resistance equivalent to 7.5% of the participant's body weight. Sprint duration will be 10 s in week 1, 15 s in week 2, and 20 s in the remaining 4 weeks. The first sprint will finish at 2 min and the second sprint will finish at 6 min. Participants will be instructed to start pedalling as fast as they can ~2-3 s before applying the sprint resistance, and to keep pedalling as fast as they can during the sprint. Verbal encouragement will be provided. Heart rate and power output will be measured throughout each 10-minute exercise session. The post-training V̇O2max test will be scheduled 3 days following the last training session.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Sedentary or recreationally active

Exclusion Criteria:

* Classified as highly physically active on the International Physical Activity Questionnaire (IPAQ)
* Answering 'Yes' to any of the questions of a standard Physical Activity Readiness Questionnaire (PAR-Q)
* Resting heart rate >100 bpm
* Resting blood pressure > 140/90 mm Hg
* BMI > 35 kg/m2
* Testing positive for Covid-19
* Pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in maximal aerobic capacity (VO2max) | Pre-intervention and 3 days following completion of the intervention.
  VO2max is the greatest volume of oxygen an individual can consume per minute. It is a key health marker.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University of Stirling, Stirling, Stirlingshire
  - University of Worcester, Worcester, Worcestershire
  - Swansea University, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD can be provided to other researchers on request, if the data are of use to answer a valid research question.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of data collection.